CLINICAL TRIAL: NCT05540821
Title: Efficacy of Double Contrast-enhanced Ultrasound of Pelvic in Preoperative Evaluation of Deep Endometriosis: a Prospective Diagnostic Test
Brief Title: Efficacy of Double Contrast-enhanced Ultrasound of Pelvic in Preoperative Evaluation of Deep Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20223357017
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Deep Endometriosis
Keywords: Deep endometriosis; contrast-enhanced ultrasound; #Enzian classification; preoperative evaluation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- conventional transvaginal ultrasound group
- double contrast-enhanced ultrasound group: perfromed hysterosalpingo-contrast sonography and sonoPODography examination
  Interventions: Diagnostic Test: Hysterosalpingo-contrast sonography and sonoPODography

INTERVENTIONS:
Diagnostic Test: Hysterosalpingo-contrast sonography and sonoPODography — Before operation, phloroglucinol 40mg of antispasmolysis was injected intramuscular, and then cervical dilation was performed according to aseptic operation requirements. A 12G double-lumen catheter was inserted into the uterine cavity, and 1.5-1.8ml of normal saline was injected into the sacculus.
  Transvaginal 2/3/4D hysterosalpingo-contrast sonography: One operator extracted 2ml of Sonovue and injected 18ml of normal saline through a dual-lumen catheter, and the other operator started the four-dimensional ultrasound mode to collect dynamic volume data.
  sonoPODography: Sterile saline was injected into the intrauterine cavity, with an upper limit of 20ml. The normal saline flowed from the intrauterine cavity into the pelvic cavity through the bilateral fallopian tubes, forming a good acoustic window. Pelvic observation was then performed.
  Groups: double contrast-enhanced ultrasound group

SUMMARY:
Endometriosis occurs in about 10-15% of women of childbearing age and is a major cause of infertility and dysmenorrhea. Deep endometriosis is the most serious manifestation of endometriosis, which often affects the quality of life of patients and requires surgical treatment. Detailed description of DE lesions before operation can contribute to treatment planning. However, the detection rate of DE by conventional ultrasound is low, highly dependent on the experience of the examiner and poor reproducibility. Hysterosalpingo-contrast sonography can be used to assess the patency of the fallopian tube but cannot visualize other pelvic structures. Saline-infusion sonoPODography can provide a good acoustic window for pelvic tissue visualization. Therefore, this study is the first to present double contrast-enhanced ultrasound (Hysterosalpingo-contrast sonography and sonoPODography) examination of the pelvic cavity, based on the #Enzian classification system, for preoperative evaluation of DE lesions. The results of laparoscopic surgery were taken as the gold standard to compare the diagnostic efficacy of double contrast-enhanced ultrasound and conventional transvaginal ultrasound in preoperative evaluation of pelvic DE lesions, improving the preoperative diagnosis, reduce the risk of surgery and reduce postoperative recurrence. To compare the diagnostic efficacy of different examination methods in different compartment of DE, and to explore the best examination method suitable for different parts of DE, providing theoretical basis for further early screening and personalized treatment of DE in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients diagnosed with adenomyosis and/or chocolate cysts, suspected infertility with endometriosis, and proposed for laparoscopic surgery at our hospital.
2. Sexual life history.
3. Surgery was performed within 2 months of the examination.
4. Subjects volunteered to participate in the study and signed the informed consent form.

Exclusion Criteria:

1. colporrhagia.
2. Acute inflammation of reproductive system.
3. Allergic to ultrasound contrast agent (Sonovue).
4. Suspected malignant lesions of cervix or uterine cavity.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consecutive female patients admitted to Shenzhen Second People's Hospital planned to undergo laparoscopic surgery from June 2022 to October 2024 with adenomyosis and/or chocolate cyst, suspected infertility complicated with endometriosis were included.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
True positive rate | Surgery was performed within 2 months of the examination
  According to the #Enzian classification system, the proportion of the number of DE lesions found by double contrast-enhanced ultrasound (DCEUS) in the pelvic cavity to the number of DE lesions found by laparoscopy.
True negative rate | Surgery was performed within 2 months of the examination
  According to the #Enzian classification system, the proportion of pelvic normal numbers shown by DCEUS to the number of pelvic normal numbers show by laparoscopy.
False negative rate | Surgery was performed within 2 months of the examination
  According to the #Enzian classification system, the proportion of pelvic DE lesions that were not detected by DCEUS in pelvic DE lesions.
False positive rate | Surgery was performed within 2 months of the examination
  According to the #Enzian classification system, in the non-pelvic DE lesions, the proportion of the number of DE lesions diagnosed by pelvic dual contrast-enhanced ultrasound accounted for.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Chen, Study Director — Shenzhen Second People's Hospital
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 1 years after publication

REFERENCES:
- [Background] Taylor HS, Kotlyar AM, Flores VA. Endometriosis is a chronic systemic disease: clinical challenges and novel innovations. Lancet. 2021 Feb 27;397(10276):839-852. doi: 10.1016/S0140-6736(21)00389-5. PMID 33640070
- [Background] Nisenblat V, Bossuyt PM, Farquhar C, Johnson N, Hull ML. Imaging modalities for the non-invasive diagnosis of endometriosis. Cochrane Database Syst Rev. 2016 Feb 26;2(2):CD009591. doi: 10.1002/14651858.CD009591.pub2. PMID 26919512
- [Background] Tuttlies F, Keckstein J, Ulrich U, Possover M, Schweppe KW, Wustlich M, Buchweitz O, Greb R, Kandolf O, Mangold R, Masetti W, Neis K, Rauter G, Reeka N, Richter O, Schindler AE, Sillem M, Terruhn V, Tinneberg HR. [ENZIAN-score, a classification of deep infiltrating endometriosis]. Zentralbl Gynakol. 2005 Oct;127(5):275-81. doi: 10.1055/s-2005-836904. German. PMID 16195969
- [Background] Exacoustos C, Malzoni M, Di Giovanni A, Lazzeri L, Tosti C, Petraglia F, Zupi E. Ultrasound mapping system for the surgical management of deep infiltrating endometriosis. Fertil Steril. 2014 Jul;102(1):143-150.e2. doi: 10.1016/j.fertnstert.2014.03.043. Epub 2014 Apr 29. PMID 24794315
- [Background] Leonardi M, Espada M, Lu C, Stamatopoulos N, Condous G. A Novel Ultrasound Technique Called Saline Infusion SonoPODography to Visualize and Understand the Pouch of Douglas and Posterior Compartment Contents: A Feasibility Study. J Ultrasound Med. 2019 Dec;38(12):3301-3309. doi: 10.1002/jum.15022. Epub 2019 May 15. PMID 31090229